CLINICAL TRIAL: NCT01222455
Title: An Open-label, Single-center Study to Assess the Pharmacokinetics of R406 in Subjects With Hepatic Impairment and in Healthy Subjects Following Administration of a Single Dose of Fostamatinib Disodium 150 mg
Brief Title: A Study of Fostamatinib in Subjects With Impaired Hepatic (Liver) Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Mark Layton / MD, AstraZeneca Pharmaceuticals
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: D4300C00010
Record Dates: First submitted 2010-10-15; First posted 2010-10-18 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2011-07

CONDITIONS: Hepatic Impairment; Healthy Volunteers; Pharmacokinetics; Amount of R406 in Blood
Keywords: Phase 1; Healthy volunteers; Volunteers with hepatic impairment; Pharmacokinetics; Fostamatinib
MeSH Terms: interventions — fostamatinib

ARMS (4):
- 1 (Experimental): Mild hepatic impairment
  Interventions: Drug: Fostamatinib
- 2 (Experimental): Moderate hepatic impairment
  Interventions: Drug: Fostamatinib
- 3 (Experimental): Severe hepatic impairment
  Interventions: Drug: Fostamatinib
- 4 (Experimental): Matched healthy volunteers with normal hepatic function
  Interventions: Drug: Fostamatinib

INTERVENTIONS:
Drug: Fostamatinib — Oral tablets, single dose

SUMMARY:
A study to evaluate the amount of fostamatinib in the blood in subjects with impaired hepatic (liver) function compared with healthy volunteers with normal liver function. The study will also evaluate safety and tolerability in subjects with hepatic impairment.

ELIGIBILITY:
Inclusion Criteria:

* Males and females (non child-bearing potential) aged 18 years or more, with a weight of at least 50 kg and body mass index (BMI) between 18 and 40 kg/m2 inclusive
* Healthy subjects only: good health as determined by a medical history, physical examination , ECG and clinical laboratory evaluations
* Healthy subjects only: negative results for serum hepatitis B and C

Exclusion Criteria:

* Subjects who have received any medications known to alter drug absorption or elimination within 30 days of first dose.
* Subjects who smoke more than 10 cigarettes or equivalent per day
* Absolute neutrophil count <2500/mm3
* Abnormal vital signs, additional systemic disease (eg, cardiac, or renal disease) or abnormal laboratory findings that are judged to be clinically significant by the investigator
* Healthy volunteers only: use of prescribed medications within 2 weeks of first dose or use of non-prescribed medications within 1 week of first dose
* Hepatic subjects only: fluctuating or rapidly deteriorating hepatic function

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2010-10; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
To determine plasma PK parameters of R406 in subjects with varying degrees of hepatic impairment as well as in healthy subjects (including but not limited to: AUC, tmax, Cmax and terminal elimination half life (t1/2)) | From pre-dose until 120 hours after the single dose

SECONDARY OUTCOMES:
To investigate safety and tolerability of fostamatinib 150mg: adverse event monitoring, vital signs, physical examinations, clinical laboratory tests, ECGs. | From pre-dose until 120 hours after the single dose

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Marbury, MD, Principal Investigator — Orlando Clinical Research Center
Locations (1):
- Research Site, Orlando, Florida, United States

REFERENCES:
- [Derived] Martin P, Oliver S, Gillen M, Marbury T, Millson D. Pharmacokinetic Properties of Fostamatinib in Patients With Renal or Hepatic Impairment: Results From 2 Phase I Clinical Studies. Clin Ther. 2015 Dec 1;37(12):2823-36. doi: 10.1016/j.clinthera.2015.09.016. Epub 2015 Oct 27. PMID 26519231